CLINICAL TRIAL: NCT01804088
Title: Clinical Investigation of the Cook Formula™ 535 Iliac Balloon-Expandable Stent
Brief Title: FORMAT Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-023
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Symptomatic Vascular Disease of the Iliac Arteries
Keywords: Peripheral artery disease; Iliac arteries; Balloon-expandable stent
MeSH Terms: conditions — Peripheral Arterial Disease

ARMS (1):
- Stent (Experimental)
  Interventions: Device: Formula™ 535 Iliac Balloon-Expandable Stent

INTERVENTIONS:
Device: Formula™ 535 Iliac Balloon-Expandable Stent — Treatment of symptomatic vascular disease of the iliac arteries

SUMMARY:
The FORMAT Clinical Study is a clinical trial to evaluate the safety and effectiveness of the Formula™ 535 Iliac Balloon-Expandable Stent in treatment of symptomatic vascular disease of the iliac arteries.

ELIGIBILITY:
Inclusion Criteria:

* Up to two documented common or external iliac artery lesions (one on each side), with >50% diameter stenosis, suitable for stenting
* iliac artery reference vessel diameter of 5-10 mm
* Rutherford Category 1, 2, 3, or 4.

Exclusion Criteria:

* Less than 18 years of age
* lesion site <10 or >100 mm in length
* external iliac artery lesion visually estimated to be 100% occluded
* presence of infrarenal aortic aneurysm >4 cm (treated or untreated)
* presence of any aneurysm (treated or untreated) within target vessel
* significant stenosis (>50%) or occlusion of inflow tract (infrarenal aortic lesions) not successfully treated before this procedure (success is measured as < 30% residual stenosis)
* absence of at least one patent runoff vessel with ≤ 50% stenosis throughout its course (i.e., confirmed in-line patency to the level of the foot)
* angiographically evident thrombus within the target vessel (treated or untreated)
* lesion is in an iliac artery that has been previously stented

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-03; Primary Completion 2015-04 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Freedom from major adverse events | 9 months

SECONDARY OUTCOMES:
Rate of technical success (i.e., successful delivery and deployment of a Formula™ 535 Iliac Balloon-Expandable Stent) | Intraoperative
Rate of acute procedure success(i.e.,vessel with <30% residual stenosis determined angiographically immediately after stent placement and no major clinical events) | Postoperative until discharge (i.e., 0 to 4 days)
Rate of hemodynamic success(i.e., ABI or TBI improved above baseline) | 30 day, 9 month, 2 year, 3 year
30-day clinical success (i.e., vessel with <30% residual stenosis determined angiographically immediately after stent placement and no major clinical events) | 30 day
Rate of primary patency (i.e.,the proportion of patients, over time, that have had uninterrupted patency since the initial procedure) | 30 day, 9 month, 2 year, 3 year
Rate of functional status improvement based on walking impairment questionnaire | 30 day, 9 month, 2 year, 3 year
Rate of improvement in Rutherford Category (i.e., improvement above baseline) | 30 day, 9 month, 2 year, 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. Geraghty, MD, Principal Investigator — Washington University School of Medicine
Locations (12):
- United States (12):
  - Scripps Health, La Jolla, California
  - CardioVascular Solutions Institute, Bradenton, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Coastal Vascular and Interventional, Pensacola, Florida
  - Peoria Radiology Associates, Peoria, Illinois
  - Indiana University Health - Methodist Hospital, Indianapolis, Indiana
  - University of Louisville, Louisville, Kentucky
  - New York-Presbyterian/Weill Cornell Medical Center, New York, New York
  - Wake Heart Research (Rex Hospital), Raleigh, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Wellmont Holston Valley Medical Center, Kingsport, Tennessee